### Title of study:

# Ward AdmiSsion of Haematuria: an Observational mUlticentre sTudy (WASHOUT)

[Study Protocol]

Protocol NCT number:

**Awaiting** 

Version:

V1.00 (Version for submission of peer review and protocol publication)

Date uploaded to clinicaltrials.gov:

19/03/2025

# A study protocol on the Ward AdmiSsion of Haematuria: an Observational mUlticentre sTudy (WASHOUT)

Nikita R.Bhatt and Kevin Byrnes (joint first), Simona Ippoliti, Raghav Varma, Bing Jie Chow, Quentin Mak, Nikki Kerdegari, Aqua Asif, Arjun Nathan, Alex Ng, Maria Ribal, John McGrath, Ben Lamb, Jim Catto, Ben Challacombe, Graeme Maclennan, Kevin Gallagher, Sinan Khadhouri, Veeru Kasivisvanathan

#### **Corresponding author:**

Veeru Kasivisvanathan, University College Hospital, University College London Hospitals NHS Foundation Trust, London, UK. veeru.kasi@ucl.ac.uk

Keywords: emergency haematuria; inpatient haematuria; clot retention; collaborative study; radiation cystitis;

#### **Abstract**

#### Introduction

Haematuria contributes significantly to emergency urology admissions. Despite over 25,000 annual UK admissions, with 10% readmitted within 30 days, there is limited focus on optimising inpatient pathways internationally. Existing studies highlight a substantial underlying malignancy rate (32%) in patients presenting with visible haematuria, yet many receive inconsistent care, leading to prolonged hospital stays and increased resource use. A systematic review (PROSPERO CRD42023466710) performed by our research group found no large-scale prospective studies have been performed in this area, and little is known about current practice. This study aims to address these gaps by investigating current management practices and their impact on outcomes, with the goal of informing evidence-based guidelines and improving patient care.

#### Methods and analysis

The WASHOUT study is an international, multicentre prospective observational study designed to describe the management of patients with unplanned admission to hospital with haematuria. The study will utilise a collaborative methodology using the BURST model. Data on demographics, comorbidities, management practices, and outcomes will be collected using a standardised case report form and analysed using multilevel linear regression modelling. Primary outcomes include length of stay, while secondary outcomes cover diagnosis time, 90-day mortality, readmission rates, and resource use. Patient and public involvement has been integral to the study design, ensuring that outcomes reflect patient priorities and that the research addresses key areas of concern.

#### **Ethics and dissemination**

Ethical and regulatory approvals will be obtained as required in each participating region. In the UK, the

study is classified as a service evaluation and does not require individual patient consent. Participating sites must obtain local audit department approval. Data will be collected and stored securely, ensuring patient confidentiality. Results will be disseminated through scientific conferences, peer-reviewed publications, and patient advocacy groups.

#### **Strengths and Limitations**

- 1. The large international, multicentre prospective study design captures real-world clinical practice, enhancing the generalizability of findings due to the diversity of data.
- 2. Broad inclusion and exclusion criteria ensure the study captures a wide variety of haematuria presentations, enabling comprehensive analysis and robust subgroup analysis.
- 3. The collaborative model of data collection, proven successful in previous studies, ensures high-quality, standardized data and sufficient power through large patient recruitment.
- 4. Patient and public involvement in the study design ensures that the research addresses relevant clinical outcomes and aligns with patient priorities, increasing the relevance and impact of the findings.
- 5. Limitations include variability in data quality across different sites, the lack of a standardized workup and management pathway, and the observational design, which limits the ability to establish causality.

#### Introduction

Over 25,000 patients are admitted each year in the UK with haematuria, contributing to at least 15% of all emergency urology admissions [1,2]. Up to 10% of these patients are readmitted with the same presentation within 30 days — patients frequently lack a durable treatment response or do not receive definitive diagnosis or management on initial presentation [2]. Despite the prevalence of this presentation, little focus has been placed on optimising inpatient pathways at a national level and reducing unnecessary resource use.

Findings from the prospective The Investigation and Detection of urological Neoplasia in paTlents referred with suspected urinary tract cancer: A multicentre analysis (IDENTIFY) study (by the BURST research collaborative) of 11,059 patients showed that 32% of patients presenting with visible haematuria had an underlying malignancy [3]. Of the remaining cohort, 40% had benign aetiology (e.g. comprising one or more of: urinary tract infections (28%), urolithiasis (25%), prostatic bleeding (37%), radiation cystitis (55%) and trauma (3%). 28% had no abnormality on investigation. Similar findings were reported by two further authors: a third of the patients presenting as an emergency with haematuria had malignancy with the rate increasing in patients with clots, while a malignancy rate of 39% was reported in a French study in patients presenting an emergency with haematuria [4,5]. More advanced bladder tumours are more likely to present as emergencies. In National Cancer Registration and Analysis Service (NCRAS) data, the rates of emergency admission for bladder cancer increased from T1 (7%) and T2/3 (16-19%) to T4 (31%) [6]. Patients in this cohort are typically elderly and frail, with multiple comorbidities and poor performance status. This cohort of patients has a high all-cause mortality rate, with a 30-day mortality rate of 5% and a one-year mortality rate of 23% [2]. Severe haematuria is often complicated by concomitant comorbidities such as cardiac failure, renal failure, history of thromboembolic events, and use of antiplatelet or anticoagulant medications [7].

In addition to poor clinical outcomes, patients admitted with haematuria require a higher resource use in terms of nursing and medical input, irrigation requirements, long inpatient stays and high readmission rates. A recent retrospective study (of 56 patients) in Ireland examining resource use associated with radiation cystitis conservatively estimated a cost burden of €23,706 per inpatient stay [8]. Radiation cystitis accounted for 621 inpatient bed days, averaging 11 days per patient. A small minority of patients are resource-intensive, some being transfusion-dependent with long inpatient stays and multiple procedures. The median length of stay for patients admitted with haematuria has increased from 8.5 days to 10 days over the last 5 years [9]. The reason behind this trend is currently unknown. This trend is the reverse of contemporary management goals such as length of stay in elective urological surgery (e.g. TURP/TURBT), for which a move toward day-case surgery (and same day of surgery discharge) has reduced unnecessary inpatient days in patients with postoperative haematuria [10].

Components of an effective inpatient haematuria pathway could potentially include specialist urology input at the point of presentation (to perform catheterisation and washout), timely imaging studies, theatre staff competent in supporting endoscopic urology, decisive intervention, consultant involvement

in operative management, acceptance of operative risk, and the avoidance of deferral to elective lists for definitive management. However, these elements of a haematuria pathway remain to be be investigated. It remains unclear which elements of management pathways are associated with best outcomes. There is a need to protocolise inpatient haematuria management in line with recommendations in other areas by Getting it Right First Time (GIRFT) national programmes.

A systematic review (PROSPERO CRD42023466710) performed by our research group found no large-scale prospective studies have been performed in this area, and little is known about current practice. Several fundamental questions about variation in practice across the UK and internationally remain unanswered including: i) What proportion of patients have a known underlying urological diagnosis? ii) What proportion of patients receive a new definitive diagnosis on index admission? iii) What proportion of patients undergo intervention during the admission? iv) Is early intervention associated with lower resource use or decreased readmission rates? v) What is the all-cause mortality in this patient cohort? vi) What proportion of patients are deemed palliative during their initial admission? vii) What proportion of patients are readmitted with the same issue? Answering these questions is essential to informing areas of best practice in this area as well as creating future research priorities for prevention and management of haematuria. The evidence available comprises small-single centre retrospective audits [2,8] evaluating mortality, readmission and cost burden of this presentation.

There are no evidence-based guideline recommendations on the timing of investigations and interventions for inpatients with haematuria. Consequently, the management of visible haematuria is currently suspected to be highly variable, both nationally and internationally but further evidence is necessary to substantiate this. Clear guidelines and standardised management pathways may reduce variability in the management of these patients. There is an urgent need to provide good quality evidence in this under-researched area to potentially improve outcomes.

#### Methods and analysis

#### Study design and aim

WASHOUT is an international, multicentre prospective observational study aiming to describe the management of patients with unplanned admission to hospital with haematuria.

#### **Objectives:**

Our objectives are:

- Establish the prevalence of causative diagnoses in patients with unplanned admission to hospital because of haematuria.
- Describe demographics, comorbidities, management, and clinical outcomes of patients with unplanned admission to hospital because of haematuria.
- Identify factors associated with adverse outcomes and/or increased resource use in this population.

- Identify if variation in management and outcomes exists at local, regional and international levels.
- Describe the impact different management pathways have on clinical outcomes (in terms of length of stay, health resource utilisation, readmission, 30-day and 90-day mortality rates.
- Provide information to design a future randomised trial, for example control group outcomes and estimates of inter-cluster correlations.

#### **Hypothesis**

The study hypothesis is that there is significant international and national variation in the diagnostic workup and management of patients requiring admission to hospital with haematuria.

Increased length of stay and poor outcomes in terms of mortality and healthcare costs are associated with clinical management practices.

#### Eligibility

#### **Patient Inclusion criteria**

Patients will be included consecutively if they are over 18 years of age and have an unplanned admission to a participating secondary care centre under the primary or joint care of the urology team due to haematuria.

In the UK, individual consent is not necessary as this study has been considered a service evaluation.

#### **Patient Exclusion criteria**

We will exclude any patients with trauma as a cause of haematuria (including catheter related trauma: defined as haematuria immediately after insertion of a urethral catheter without a preceding history of haematuria on this admission including traumatic catheter removal by patients), urological trauma (abdominal/pelvic) as well as patients who are in hospital less than 24 hours. Our study steering group felt this population had several confounders, including inappropriate admissions. Including these patients would mix the study population with patients best served by outpatient investigation and management (for which guidelines currently exist to guide practice)

#### Site inclusion criteria

Secondary care centre with a urology-specific unit/ team that accepts unplanned admissions anywhere in the world.

#### Site exclusion criteria

Sites lacking a minimum standard of data quality and completion will be excluded

#### Outcomes

As WP1 lacks an experimental design; it is not powered to a specific primary outcome. However, to emulate outcomes of interest for a target trial in WP3 we identified primary and secondary outcomes with public and patient involvement.

#### **Primary outcome**

Length of stay (LoS), measured in calendar days. A basic definition of LoS is the number of days measured as an integer by taking the date of admission in the index hospital admission episode and the date of discharge from the hospital, and calculating the date difference between them. Variations in exact definitions of length of stay will be reported. Examples of this are including calendar days spent in the emergency department, or excluding days after care of the patient is taken over by another team, or after being medically discharged.

#### **Secondary outcomes**

- For those without a previously known cause of haematuria: time to definitive diagnosis, defined as the number of days between original presentation and final diagnosis.
- Length of time required to be in hospital for hospital, measured as an integer by taking the date of admission in the index hospital admission episode and the date of discharge from the hospital or the date deemed medically fit for discharge (whichever is first), and calculating the date difference between them.
- 90-day mortality rate measured as the proportion of patients who died from the day of admission to the 90-day follow-up period.
- 90-day readmission rate, measured as the proportion of patients who were readmitted to the hospital with the same issue in the 90-day after the date of discharge.
- Number of days alive and out of hospital at 90 days.
- Resource use, including inpatient days and investigations and procedures that the patient underwent during the admission and in the 90-day follow-up period.
- The study will also assess current pathways that exist in hospitals, including acute care pathways and specific pathways for management of haematuria. Details will be obtained through a questionnaire distributed to each participating site.

#### Sub-group analysis

- Plan to report outcomes of study for the following diagnostic sub-groups:
  - Radiation cystitis
  - Urological malignancy (including pre-existing and new diagnoses)
  - Unknown diagnosis at presentation

#### Study setting

This study will take place in urological secondary and tertiary care centres internationally. The study will be conducted in centres that agree to participate in the study and meet the study's inclusion criteria below.

#### Study delivery

The study will utilise the The British Urology Researchers in Surgical Training (BURST) collaborative model which has been previously applied to observational studies globally [11]. In IDENTIFY, we recruited 11,029 patients to a multicenter observational study [3]. RESECT an observational, international, multicenter study with an embedded cluster randomised trial of audit, feedback, and education and recruited 19,500 cases[12]. The design of the current study has been supported by input from the Centre for Healthcare Randomised Trials (CHaRT) (i.e. The Urology Foundation trials unit), who will be involved in designing and conducting the next study, which we anticipate will be an implementation randomised controlled trial.

#### Recruitment

Patients will be recruited consecutively. The recruitment target for this study is based pragmatically on the prevalence of inpatient haematuria. Target recruitment per participating site is 15 patients across a 12-month period from 70 centres. The cumulative recruitment target from all sites is 1,050 patients. We want to recruit as many participants as possible during the 12-month period. The sample size is also based on the anticipated wide variation of practice and the heterogeneous nature of the presentation in terms of patient demographics and the underlying cause of the haematuria ranging from benign causes to malignant urological conditions [1, 2].

This sample size is also adequately powered to detect a meaningful difference in length of stay (defined as at least 1 day by study authors) using ANOVA to analyse any binary variable (spanning both clinicopathological features and management factors). This 1-day difference in length of stay is based on a calculated sample size of 1,054 patients, obtaining a power of 0.90 with a significance level of 0.05, and taking a standard deviation of length of stay as 5 days obtained from original data of a retrospective review covering this study population [2].

#### **Data collection**

Participating sites will complete a registration survey describing their institution and urological practice (sub-specialities and consultants, on-call rota and support) and if any local protocols or defined criteria for referral/admission exist - Appendix 2).

Data will be collected prospectively on consecutive patients requiring emergency admission over a 12-month period. Non-identifiable patient data will be collected by individual investigators using the REDCap electronic data capture tool. Data will be collected prospectively by the participating centres using a standardised case report form (CRF). The CRF will include data on demographics, medical history, aetiology of haematuria, length of stay, investigations, interventions, complications, health resource utilisation, readmissions, and 30-day and 90-day mortality rates. Data will also be collected on

interventions (if any) including ward management, surgical, radiological and any other interventions or adjunct treatments. Data collected is information recorded as part of clinical assessment, thereby allowing local sites to qualify as a process evaluation in the UK setting. Further details are available in Appendix 1 and 2.

Data will be entered into a secure online UCL Redcap database. All data collected will be kept confidential and anonymous. Each participating centre will be assigned a unique identifier code, and no personal identifying information will be collected from the patient or managing surgeon. Where available, standardised clinical data models will be used to structure data collection. We will ensure each site has registered with the relevant local audit department that they are undertaking an evaluation of current practice.

#### **Data analysis**

We will describe the cohort demographic and clinical variables at baseline, using descriptive statistics.

We will use multilevel linear regression modelling to analyse primary outcome length of stay (LoS) to understand the variation across centres, extending this to model the association between LoS and factors such as age, gender, comorbidities, and management practices. Missing data will be handled using multiple imputation and pattern mixture models. Secondary outcomes will be analysed similarly using the appropriate multilevel generalised linear model for the distribution of the outcome.

Descriptive resource use information will be presented according to standard categories, and standard unit costs (NHS Reference Costs) applied where appropriate to provide information on costs of the observed patient diagnostic and therapeutic pathways.

#### Patients who do not complete follow-up period

Investigators who enter a follow-up period earlier than 90 days will be included in the analysis for the outcomes of length of stay, readmission and mortality. Resource use will be included if entered in the 15 days prior to 90 day follow-up or any point after.

#### **Ethics and dissemination**

Before beginning the study, ethical and local regulatory approval as required in each respective region, will be obtained in accordance with applicable guidelines. In the UK, the Health Research Authority and the National Research Ethics Service advised that this study was exempt from ethical approval. The letter supporting this is attached as Appendix 3. Each participating UK site will require approval from their local audit department and/or research and development office. The international sites will be provided with study documentation to apply for local ethics approval.

Once the study is complete, the results will be presented at international scientific conferences in the field of urology, published in peer-reviewed journals, and shared with patient advocacy groups via Urology charities, including the Urology Foundation (TUF), the European Association of Urology patient

office and our patient and public involvement (PPI) panel. We are committed to ensuring that all collaborators who make significant contributions to the study will be listed as collaborative authors on Pubmed-indexed papers resulting from the study as per the BURST authorship policy used in previous BURST projects [9]. We will communicate findings to leading associations, including NICE and EAU. We will also disseminate research findings using different (social) media platforms.

#### **Quality control**

An independent quality control team will thoroughly check all data submitted to ensure accuracy and completeness. Incomplete or outlier data will be identified, and investigators will be contacted to address any issues.

#### **Patient Public Involvement**

A total of 10-15 patients who have been admitted with haematuria were identified by directly contacting patients admitted to hospital with this condition, marketing through social media and patient focus groups as well as charities. Anyone with a personal experience of blood in their urine requiring hospital admission or a relative or friend of a patient suffering from this condition was eligible as a patient representative. Public representatives could include lay members of the public with an interest in patient improvement research. Ethics was not necessary as this was deemed as involvement work and feedback on study design was collected rather than any study data. They were invited to a virtual meeting on Zoom to explore outcomes of interest, aspects of care that they deem important, and identify areas of satisfaction or dissatisfaction within the management pathway. The PPI panel were remunerated for their time and input.

During the first PPI group meeting, a BURST committee member introduced the study, providing an overview of its objectives and expected outcomes. The meeting was coordinated by a PPI facilitator based in the University College of London (UCL). Participants shared their personal experiences with haematuria, discussing symptoms, diagnosis, and the impact on their lives. Patients were briefed on the study's objectives, design, and research methods, seeking their input on study parameters via an open discussion during the meeting and via a 10-item questionnaire sent via email. Patients and researchers reviewed the potential benefits and risks of the study, highlighting any concerns or suggestions.

#### The focus group agreed that:

- > The study is both valuable and they would prefer a standardised pathway for haematuria management following emergency hospital admission
- No concerns were expressed regarding the study
- The study primary and secondary outcomes (e.g.: length of hospital admission, 30-day and 3-month mortality rate, readmission rate and resource utilisation) are important to patients
- ➤ Care should be taken to create a standardised pathway which includes a prompt management of the patients when presenting symptoms of clot retention in the emergency department or in the community (e.g.: by promoting fast-track to specialty or access to adequate points of care).

As a result of PPI involvement, changes have been made to the case report form on aspects of ward management as patients felt this was important. Specifically, they expressed getting prompt access to catheterisation, washouts and irrigation was important.

#### **References:**

- [1] Hospital Episode Statistics, Hospital Admitted Patient Care Activity. NHS Digital. 2022.https://digital.nhs.uk/data-and-information/data-tools-and-services/data-services/hospital-episode-statistics (accessed January 1, 2022).
- [2] Pavithran A, Bhatt NR, Banerjee G, Hawizy A. Management of Inpatient Macroscopic Haematuria: A Typical Urology Emergency with a High Mortality. Urology 2022;166:22–8.
- [3] Khadhouri S, Gallagher KM, MacKenzie KR, Shah TT, Gao C, Moore S, et al. The IDENTIFY Study: The Investigation and Detection of Urological Neoplasia in Patients Referred with Suspected Urinary Tract Cancer; A multicentre observational study 2021.
- [4] Gan J, Harris A, Green J. Quantifying the risk of malignancy in patients with visible haematuria presenting to the emergency department. Journal of Clinical Urology. 2015;8(2):132-138. doi:10.1177/2051415814548913
- [5] Errando Smet C, Martinez De Hurtado J, Regalado Pareja R, Huguet Pérez J, Montlleó Gonzalez M, López Duesa L, Bakali Mourabet K, Chéchile Toniolo G, Vicente Rodriguez J. Analyse de 895 consultations pour hématurie dans le département des urgences d'un service d'urologie [Analysis of 895 consultations for hematuria in the emergency department in an urology unit]. J Urol (Paris). 1996;102(4):168-71. French. PMID: 9091567.
- [6] Catto JWF, Mandrik O, Quayle LA, Hussain SA, McGrath J, Cresswell, J, Birtle AJ, Jones RJ, Mariappan P, Makaroff LE, Knight A, Mostafid H, Chilcott J, Sasieni P, Cumberbatch M. Diagnosis, treatment and survival from bladder, upper urinary tract, and urethral cancers: real-world findings from NHS England between 2013 and 2019. BJU Int. 2023 Jun;131(6):734-744. doi: 10.1111/bju.15970. Epub 2023 Feb 7. PMID: 36680312.
- [7] Satasivam P, Reeves F, Lin M, Daruwalla J, Casan J, Lim C, et al. The effect of oral anticoagulation on the prevalence and management of haematuria in a contemporary Australian patient cohort. BJU Int 2012;110:80–4.
- [8] Gilmartin B, O' Meara SO, D'arcy FTD, Dowling CMD. A0083 Cost burden of radiation cystitis presentations and investigations to a tertiary referral hospital in Ireland. Eur Urol 2023;83:S122. <a href="https://doi.org/https://doi.org/10.1016/S0302-2838(23)00140-9">https://doi.org/https://doi.org/10.1016/S0302-2838(23)00140-9</a>.
- [9] NHSE. GIRFT All Clinical Metrics [Internet]. Model Health System Website. 2023 [cited 2023 Apr 18]. Available from: https://model.nhs.uk/home
- [10] Gray WK, Day J, Briggs TWR, Harrison S. Transurethral resection of bladder tumour as day-case surgery: Evidence of effectiveness from the UK Getting it Right First Time (GIRFT) programme. J Clin Urol 2020;13:221–7.
- [11] Kasivisvanathan V, Ahmed H, Cashman S, Challacombe B, Emberton M, Gao C, et al. The British Urology Researchers in Surgical Training (BURST) Research Collaborative: an alternative research model for carrying out large scale multi-centre urological studies. BJU Int 2018;121. https://doi.org/10.1111/bju.14040.

[12] Wang B, Gallagher K, Bhatt N, Clement K, Zimmermann E, Khadhouri S, et al. MP08-10 GLOBAL VARIATION IN EARLY RECURRENCE AFTER TRANSURETHRAL RESECTION OF BLADDER TUMOR IN THE RESECT STUDY (NCT05154084): THERE IS SIGNIFICANT INTER-SITE VARIATION THAT IS INDEPENDENT OF DIFFERENCES IN TUMOUR FACTORS. J Urol 2023;209:e97.

#### **Author contributions**

Study concept: NB, KB and VK

Study design: NB, KB, SK, KG, GM, VK

Protocol writing: NB, KB

Protocol editing and revisions: NB, KB, VK, GM, SI, RV, NK, BC, QM, AN, AA, ANg, SK, KG, GM, MR, BC,

JM, JC, BL.

#### **Funding:**

This work was supported by

The Urology Foundation & The Charles Reynolds Foundation - Innovation and Research Award 2024 (awarded 24 May 2024)

Action Bladder Cancer UK - Improving Outcomes for Patients Programme 2024 (awarded 29 May 2024)

# Appendix 1: Variables to be collected on each patient (to be discussed with PPI group and finalised)

#### **Patient factors**

- Baseline demographic information including age, gender
- ASA grade
- Frailty index
- Antithrombotic agents (anticoagulants and antiplatelets)
- Smoking history
- Previous radiation
- Details of clinical history
- Previous urological history

#### Haematuria factors

- Reason for referral / clinical presentations of haematuria (haematuria / clot retention, pain, dysuria/cystitis, pyelonephritis/urosepsis, upper tract obstruction, re-presentation/re-admission to ED within 30 days)
- Use of blood products or reversal agents
- Use of antibiotics
- Tranexamic acid
- Transfusion rates
- Examination findings/ Initial Observations / Sepsis- DRE
- Urine microscopy results
- Blood test results during admission e.g. AKI, low Hb, coagulation issues
- Imaging timing and results during admission
- Ward based management during admission for example catheterisation, washout, irrigation
- Level of ward care (Intensive Treatment Unit/High Dependency Unit/Ward)
- Procedure results during admission e.g. rigid cystoscopy and washout, TURBT etc
- Grade of operating surgeon
- Findings at procedure
- Complications of procedure performed
- Length of stay
- Palliative care involvement
- Healthcare resource use (imaging studies performed, procedures performed)

#### Disease factors

- Underlying aetiology
- Number of previous admissions for the same reason
- Readmission rate over 30 days and 90-days
- 30-day and 90-day mortality rate
- VTE; rate of DVT/PE

## Appendix 2. Information from centres regarding current management of unscheduled haematuria admissions

- 1. Does your unit have a protocol for inpatient management of haematuria?
- 2. Are there defined admission criteria for patients presenting with visible haematuria? If so, please define these.
- 3. Describing the type of institution (district general hospital versus tertiary university hospital, academic centre/
- 4. Describe urological practice of consultants (sub-specialities and consultants)
- 5. Is the site split into emergency and elective sites?
- 6. How is care delivered/structured (who receives referrals consultant or registrar led on-call)?

- 7. Do you have bedside flexible cystoscopy available?
- 8. Is there a dedicated urology treatment room contained within the acute care component of your hospital (is it staffed by CNSs, equipment available, protocols defined).
- 9. Ward rounds led by registrar/consultant
- 10. Do you have access to same day imaging leave free text as well
- 11. Do you have access to dedicated CEPOD facilities
- 12. Do you have interventional radiology on-site
- 13. Is the primary on-call team free from elective commitments on-call
- 14. Grade of clinician accepting urology referrals during the day (consultant, reg, SHO, ANP/CNS)
- 15. Grade of clinician accepting urology referrals overnight (consultant, reg, SHO, ANP/CNS)
- 16. Do you have access to a one-stop haematuria clinic for investigating patients with haematuria?